CLINICAL TRIAL: NCT05498870
Title: Studying the Effects of iPACK Blocks With Adductor Canal Blocks for Postoperative Analgesia Following ACL Reconstruction
Brief Title: iPACK for Post-op Pain Following ACL Reconstruction
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Medical University of South Carolina (Other)
Responsible Party: Principal Investigator, Carey Brewbaker, Assistant Professor, Medical University of South Carolina
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Pro00121103
Record Dates: First submitted 2022-07-27; First posted 2022-08-12 (Actual); Results first posted 2024-07-10 (Actual); Last update posted 2024-10-16 (Actual); Status verified 2024-10

CONDITIONS: ACL Injury; Post Operative Pain
Keywords: acl injury; acl repair
MeSH Terms: conditions — Anterior Cruciate Ligament Injuries; Pain, Postoperative | interventions — Single Person

STUDY DESIGN:
Who Masked: Participant
Masking Description: Only the patient will be blinded to the treatment group.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Adductor Canal Block (ACB) Only (Active Comparator): Participants randomized to the ACB only group will receive an adductor canal block alone.
  Interventions: Drug: Adductor Canal Block (ACB) Only
- ACB + iPACK (Active Comparator): Participants randomized to the ACB + iPACK group will receive both the ACB and iPACK block.
  Interventions: Drug: Adductor Canal Block (ACB) + iPACK Block

INTERVENTIONS:
Drug: Adductor Canal Block (ACB) Only — Patients will receive an ACB with lidocaine skin wheal
  Arms: Adductor Canal Block (ACB) Only
Drug: Adductor Canal Block (ACB) + iPACK Block — Patients will receive an ACB with iPACK block
  Arms: ACB + iPACK

SUMMARY:
This study will consist of patients 12 years and older undergoing ACL reconstruction using a quadriceps or bone-patella tendon bone (BTB) graft. The patients will be randomized to adductor canal block alone, or adductor canal block + iPACK block. The primary goal will be to determine the differences in postoperative pain during the first 72 hours when comparing the two groups. Secondary outcomes will include opioid utilization during the first 72 hours postoperatively and range of motion including terminal knee extension at postoperative follow-up visits.

ELIGIBILITY:
Inclusion Criteria:

* Age 12 years and older
* Patients who are scheduled to undergo an ACL reconstruction with quadriceps or BTB graft.

Exclusion Criteria:

* Any contraindication to receiving regional anesthesia. This may include infection at the site of injection, allergy to local anesthetic, or pre-existing nerve injury.
* Patients undergoing hamstring graft or allograft for ACL
* Pre-existing infection at the site of injury
* Patients on chronic opioid treatments
* Pre-existing sensory or motor deficit in operative extremity
* Patients having a revision of previous ACL reconstruction
* Pregnant and/or lactating women
* Weighs less than 40kg

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 82 (Actual)
Dates: Start 2022-08-25 (Actual); Primary Completion 2023-07-03 (Actual); Study Completion 2023-08-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Carey Breabaker, MD, Principal Investigator — Medical University of South Carolina
Locations (1):
- Medical University of South Carolina, Charleston, South Carolina, United States

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Each participant contributed one study knee. They underwent an ACL reconstruction on one single knee to qualify for participation in the study.
Period: Overall Study
Arm/Group | Adductor Canal Block (ACB) Only | ACB + iPACK
Started | 41 | 41
Completed | 34 | 38
Not Completed | 7 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Adductor Canal Block (ACB) Only | ACB + iPACK | Total
Number analyzed (Participants) | 34 | 38 | 72
Age, Continuous [Mean (Standard Deviation); unit: years] | 22.6 (8.74) | 22.8 (8.53) | 22.7 (8.62)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 20 | 36
  Male | 18 | 18 | 36
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 1 | 3
  Not Hispanic or Latino | 32 | 37 | 69
  Unknown or Not Reported | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 24 | 27 | 51
  Black | 9 | 9 | 18
  Other | 1 | 2 | 3
Body Mass Index [Mean (Standard Deviation); unit: kg/m^2] | 25.4 (3.49) | 25.9 (5.46) | 25.7 (4.63)
Preoperative VAS Pain Score [Median (Inter-Quartile Range); unit: units on a scale] | 0 [0 to 3] | 0 [0 to 5] | 0 [0 to 4]
ACL Side [Number; unit: participants] — Left ACLs vs. Right ACLs repaired
  participants
    Left ACL | 17 | 16 | 33
    Right ACL | 17 | 22 | 39

OUTCOME MEASURES:

1. Primary Outcome: Pain Scores
Description: The primary endpoint will measure subjective pain scores using a Visual Analog Scale ranging from 0 (no pain) to 100 (severe intolerable pain) at 12-hour intervals during the first 72 hours of the postoperative window. A higher score means worse outcome.
Time Frame: 0-72 hours post op
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Adductor Canal Block (ACB) Only | ACB + iPACK
Number analyzed (Participants) | 34 | 38
units on a scale
  Pain at Discharge | 41.5 (27.3) | 29.8 (20.5)
  12 hours post-op | 37.9 (4.22) | 47.4 (4.02)
  24 hours post-op | 38.7 (4.05) | 49.9 (4.32)
  36 hours post-op | 40.9 (4.84) | 54.7 (4.35)
  48 hours post-op | 40.2 (4.66) | 50.8 (4.68)
  60 hours post-op | 41.1 (4.39) | 44.2 (4.2)
  72 hours post-op | 36.2 (4.8) | 36.7 (4.15)

2. Secondary Outcome: Total Postoperative Opioid Consumption (Total MME)
Description: The secondary endpoints will measure perioperative opioid consumption through postoperative day 2 in 12-hour intervals and converted into morphine milligram equivalents using standard conversions.
Time Frame: up to 72 hours post-op
Measure: Mean (Standard Error); unit: morphine milligram equivalents
Arm/Group | Adductor Canal Block (ACB) Only | ACB + iPACK
Number analyzed (Participants) | 34 | 38
morphine milligram equivalents
  12 hours post-op | 8.26 (1.99) | 11.2 (1.93)
  24 hours post-op | 6.09 (1.98) | 10.5 (2.05)
  36 hours post-op | 10.4 (2.48) | 16.2 (2.97)
  48 hours post-op | 6.51 (2.15) | 10.5 (2.43)
  60 hours post-op | 10.5 (2.52) | 14.5 (2.55)
  72 hours post-op | 6.65 (2.18) | 7.65 (2.66)

3. Secondary Outcome: Range of Motion (Degrees)
Description: An additional secondary endpoint is the range of motion, measured in degrees, of the operative knee at post-op visit 1 and 2. The post-op measurements will be compared to the pre-operative measurements. The scale of range of motion is from 0 - 135 degrees. The higher the score (degrees), the better the outcome.
Time Frame: up to two months after surgery
Measure: Mean (Standard Error); unit: degrees
Arm/Group | Adductor Canal Block (ACB) Only | ACB + iPACK
Number analyzed (Participants) | 34 | 38
degrees | 90.0 (2.38) | 99.3 (2.23)

ADVERSE EVENTS:
Time Frame: Adverse events were collected from the time randomization occurred through the end of post-op Day 3, an average of 4 days.
Description: Patients self reported if they developed any type of nerve-block related adverse event such as nerve damage, local anesthetic systemic toxicity (LAST), numbness, or infection at injection site, etc. Additionally, they also self-reported if they had any surgical adverse events such as incision infection. All patient-reported adverse events were followed up on to confirm reported details.
Arm/Group | Adductor Canal Block (ACB) Only | ACB + iPACK
All-Cause Mortality (participants affected / at risk) | 0/34 | 0/38
Serious Adverse Events (participants affected / at risk) | 0/34 | 0/38
Other Adverse Events (participants affected / at risk) | 6/34 | 8/38
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Adductor Canal Block (ACB) Only (N=34) | ACB + iPACK (N=38)
Nerve Block Adverse Event (Injury, poisoning and procedural complications) | 2 (2) | 3 (3) — Any event reported to be cause by the nerve block. This can include nerve damage, numbness and tingling, infection at injection site, etc.
Surgical Adverse Event (Surgical and medical procedures) | 4 (4) | 5 (5) — Adverse event related to the ACL repair. This can include infection at surgical incision site, etc.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-06-17): https://cdn.clinicaltrials.gov/large-docs/70/NCT05498870/Prot_SAP_000.pdf